CLINICAL TRIAL: NCT01687647
Title: Interest of Morphometric Analysis of Sputum Cytology for Lung Cancer Screening in Workers Highly Exposed to Asbestos - Exploratory Analysis of Biomarkers Predictive for Lung Cancer
Brief Title: Sputum Cytometry Analysis in Lung Cancer Screening After Professional Asbestos Exposure
Acronym: AMORCE-CBP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Caen (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 2011-A01380-41; PHRC11-221 (Other Grant/Funding Number: French Ministry of Health (DGOS))
Record Dates: First submitted 2012-08-31; First posted 2012-09-19 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Lung Neoplasms
Keywords: Lung cancer screening; Asbestos exposed workers; Sputum analysis; Automated cytometry; Predictive biomarkers
MeSH Terms: conditions — Lung Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening (Other): Paired-design: low-dose CT scan, sputum sample and blood test will be performed on all subjects.
  Interventions: Other: low-dose CT-scan AND induced sputum sample AND blood test

INTERVENTIONS:
Other: low-dose CT-scan AND induced sputum sample AND blood test — All subjects will receive a low-dose CT-scan, a blood test (ancillary study) and provide an induced sputum

SUMMARY:
Workers exposed to asbestos are at high risk of lung cancer. Medical follow-up of this population relies on repeated CT-scans which are more accurate for detection of peripheral lesions, and expose to X-rays and to risk of false-positives. Analysis of sputum using automate cytometry may be of interest in this population, alone or in combination with CT-scan.

An ancillary study will evaluate the interest of blood predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* High professional asbestos exposure
* Member of a former cohort recruited between 2000 and 2006 in Caen, Rouen and Le Havre (inclusion criteria: 50-75 years at the time of initial recruitment, high intermittent asbestos exposure >= 1 year, or high discontinuous asbestos exposure >=10 years). All the living members of the cohort will be contacted: a maximum of 1000 subjects is expected, probably less.
* Informed consent signed

Exclusion Criteria:

* Personal history of lung cancer
* Refusal of the study protocol
* Uncontrolled asthma or lung failure

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Risk of false positive | within 3 months
  Ratio of false positives (RFP) for detection of lung cancer in reference to conventional cytology analysis of sputum
detection of lung cancer | within 3 months
  Ratio of sensitivities for detection of lung cancer in reference to conventionnal cytology analysis of sputum

SECONDARY OUTCOMES:
Sensitivity for lung cancer detection compared with CT-scan | within 3 months
  Ratio of sensitivity (RSN) for lung cancer detection in reference with CT scan.
  Interest of the combination "cytometry + CT-scan" compared with CT-scan alone will also be evaluated.
Specificity for detection of lung cancer | within 3 months
  Ratio of false positives (RFP) of automated cytometry analysis compared with CT-scan screening.
  The combination "automated cytometry + CTscan" will also be evaluated compared with CT scan alone.
Predictive Biomarkers | Annually during a maximum of 5 years
  Frequency of specific biomarkers at the time of screening. Links between lung cancer during 5 years of prospective follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia GUITTET, MD,PhD, Study Director — Caen University Hospital, INSERM
Locations (3):
- France (3):
  - Caen University Hospital, Caen
  - Le Havre Hospital, Le Havre
  - Rouen University Hospital, Rouen